CLINICAL TRIAL: NCT01694381
Title: Phase 1 Trial of Mutant proUK, M5, and Its Inhibitor, C1-inhibitor
Brief Title: Research Into the Effect of a Clot-dissolving Agent and Its Inhibitor
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: TSI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS01-01; 2012-002225-30 (EudraCT Number)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; TS01; Mutant pro-urokinase; M5; C1 inhibitor; Safety; Stroke; Tolerability; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Brain Infarction; Brain Ischemia; Fibrinolytic Agents; Thrombolytic Agents; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Cardiovascular Agents; Therapeutic Uses; Hematologic Agents
MeSH Terms: conditions — Ischemic Stroke; Angioedemas, Hereditary; Stroke; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Brain Infarction; Brain Ischemia | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Intervention Model Description: The trial consists of two study parts in which healthy male volunteers will randomly and in a double-blinded manner receive a single dose of M5 or M5-placebo intravenously, with (part II) or without (part I) a preceding single dose of C1-inhibitor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mutant pro-urokinase (M5) alone (Experimental): In the first study part subjects in cohorts of 4 will receive ascending doses of either M5 (3 subjects) or M5-placebo (1 subject) without C1-inhibitor.
  Interventions: Drug: M5
- Mutant pro-urokinase (M5) and its inhibitor, C1 inhibitor (Experimental): In the second study part subjects in cohorts of 5 will receive ascending doses of either M5 or M5-placebo, preceded by a single intravenous dose of C1-inhibitor or C1-inhibitor-placebo. Each subject will randomly be allocated to one of the following treatment arms within one cohort:
  * C1-inhibitor followed by M5 (3 subjects);
  * C1-inhibitor followed by M5-placebo (1 subject);
  * C1-inhibitor-placebo followed by M5-placebo (1 subject).
  Dose levels of both M5 and C1-inhibitor within each cohort will be chosen based on the available safety, pharmacokinetic and pharmacodynamic data of the preceding cohorts.
  Interventions: Drug: M5; Drug: C1-inhibitor

INTERVENTIONS:
Drug: M5 — single point mutant of serine protease prourokinase
Drug: C1-inhibitor — a protease inhibitor belonging to the serpin superfamily.
  Arms: Mutant pro-urokinase (M5) and its inhibitor, C1 inhibitor

SUMMARY:
Single-chain urokinase-type plasminogen activator (pro-urokinase) is a highly effective thrombolytic drug. At pharmacologic concentrations however, pro-urokinase is converted to urokinase - a non specific thrombolytic, limiting its therapeutic use. Mutant pro-urokinase (M5) is more stable and its conversion to urokinase is inhibited by C1-inhibitor.

The primary objectives of the study are:

* To assess the overall safety and tolerability related to systemic plasminogen activation of single doses of M5 over a wide dose range (study part I).
* To assess the effect of single doses of C1-inhibitor on the overall safety and tolerability of single doses of M5 and its effect on M5-induced coagulation changes (study part II).

DETAILED DESCRIPTION:
Mutant proUK, M5, was specifically designed to improve the plasma stability of single-chain proUK by reducing its intrinsic catalytic activity and allowing it to retain its proenzyme form until it encounters a thrombus. As an additional consequence of the mutation, its two-chain enzymatic form (tcM5) is sensitive to inhibition by C1-inhibitor (C1INH) a relatively abundant plasma inhibitor.

While it has a negligible effect on urokinase (UK), C1INH inhibits tcM5 irreversibly, preventing non-specific plasminogen activation, responsible for bleeding complications. The effect of endogenous C1INH can be augmented by the addition of exogenous C1INH. In vitro studies in rats and dogs indicated that adding C1INH to plasma prior to clot lysis by M5 prevented bleeding, fibrinogenolysis and plasminogen depletion but did not affect the rate of fibrinolysis. In a recent pilot rat stroke study, at similarly effective doses, M5, preceded by C1INH adjunctive therapy, was equivalent to tPA alone but caused significantly less ICH, was much more effective than tPA preceded by adjunctive C1INH, and was the only group with a significant functional improvement at 24h.

Dose restrictions which limit efficacy of tPA-based thrombolysis are expected to be circumvented by M5 preceded by adjunctive C1INH. C1INH is a commercially available plasma derived product with a well-established safety and efficacy profile and is currently indicated and available for routine prophylaxis of hereditary angioedema (HAE).

ELIGIBILITY:
Inclusion Criteria:

* Be male, aged between 18 and 35 years inclusive, and with a body weight of at least 60 kg and a body mass index (BMI) between 18.5 and 25 kg/m2 inclusive.
* Be without clinical significant abnormalities according to the investigator's judgment, based on a detailed medical history, a complete physical examination (including vital signs), a standard 12-lead electrocardiogram, urinalysis, and routine clinical laboratory tests.
* Have endogenous C1-inhibitor, α2-antiplasmin, fibrinogen, and plasminogen levels within the laboratory's reference range.
* Have a negative serology for HIV, HBsAg, and HCV.
* Have a negative test for alcohol and drugs of abuse at screening and on study day -1.
* Be capable of understanding and willing to comply with the conditions and restrictions of the protocol.
* Have read, understood and provided written informed consent.

Exclusion Criteria:

* Has a known or suspected inherited, congenital, or acquired disease or condition that affects the haemostatic or coagulation pathways or that is associated with an increased bleeding tendency.
* Has a reasonable chance of developing a clinically significant bleeding event or a bleeding event that may go undetected for a considerable amount of time during the study, for example:
* Has undergone major (internal) surgery or trauma within the last three months of the anticipated dosing day;
* Has an intestinal or cerebral vascular malformation;
* Has participated in high impact contact sports, such as kick-boxing, within two weeks of the anticipated dosing day.
* Has received any systemically absorbed drug or substance (including prescription, over-the-counter, or alternative remedies) that is not permitted by this protocol prior to dosing without undergoing a wash-out period of at least seven times the elimination half-life of the product. For aspirin or other products inhibiting thrombocyte-aggregation the wash-out period must not be less than 28 days.
* Has smoked tobacco in any form within three months of dosing, or has ever smoked more than five cigarettes per day (or equivalent) on average.
* Has received blood or plasma derivatives in the year preceding the administration day.
* Has lost blood or plasma outside the limits of the local blood donation service (i.c. Sanquin) three months prior to dosing.
* Has a known hypersensitivity to any of the investigational material or related compounds.
* Has a history of severe hypersensitivity or of an allergy with severe reactions.
* Has a history of substance abuse, including caffeine, tobacco, and alcohol.
* Has a condition or demonstrates an attitude that in the opinion of the investigator might jeopardise the subject's health or well-being, or the scientific integrity of the study results.
* Is mentally or legally incapacitated to provide informed consent.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes to vital signs, routine safety laboratory results, or ECG-findings | -42d, -14h, -15', 15', 30', 45',60', 90', 10h, 24h, 48h, 7d

CONTACTS AND LOCATIONS:
Overall Officials: Koos Burggraaf, MD, PhD, Principal Investigator — Center for Human Drug Research
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Background] Tomasi S, Sarmientos P, Giorda G, Gurewich V, Vercelli A. Mutant prourokinase with adjunctive C1-inhibitor is an effective and safer alternative to tPA in rat stroke. PLoS One. 2011;6(7):e21999. doi: 10.1371/journal.pone.0021999. Epub 2011 Jul 14. PMID 21779364
- [Background] Pannell R, Kung W, Gurewich V. C1-inhibitor prevents non-specific plasminogen activation by a prourokinase mutant without impeding fibrin-specific fibrinolysis. J Thromb Haemost. 2007 May;5(5):1047-54. doi: 10.1111/j.1538-7836.2007.02453.x. PMID 17459007
- [Background] Gurewich V, Pannell R, Simmons-Byrd A, Sarmientos P, Liu JN, Badylak SF. Thrombolysis vs. bleeding from hemostatic sites by a prourokinase mutant compared with tissue plasminogen activator. J Thromb Haemost. 2006 Jul;4(7):1559-65. doi: 10.1111/j.1538-7836.2006.01993.x. PMID 16839354
- [Background] Liu JN, Liu JX, Liu Bf BF, Sun Z, Zuo JL, Zhang Px PX, Zhang J, Chen Yh YH, Gurewich V. Prourokinase mutant that induces highly effective clot lysis without interfering with hemostasis. Circ Res. 2002 Apr 19;90(7):757-63. doi: 10.1161/01.res.0000014825.71092.bd. PMID 11964367